CLINICAL TRIAL: NCT03841214
Title: Prediction of ST2 for impRovement of Left ventricUlar Systolic funcTion After Percutaneous Coronary Intervention in Patients With acutE Coronary synDrome
Brief Title: Study on Prediction of Left Ventricular Remodeling Using ST2
Acronym: TRUSTED
Status: Completed | Type: Observational
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Kim Hyungseop, Professor, Keimyung University Dongsan Medical Center
Other Study IDs: TRUSTED
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2020-06

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients who underwent percutaneous coronary intervention after diagnosis of acute coronary syndrome should be enrolled in the study and follow - up.

DETAILED DESCRIPTION:
Obtain written consent for patients who meet all of the selection criteria and who do not meet the exclusion criteria.

ACS(Acute Coronary Syndrome) patients with LV systolic dysfunction(LVEF<50%) on TTE test who underwent successful PCI. At that time, patient proceed with the Baseline blood test(ST2) in hospital.

And then, Medical therapy for 3 months later patient proceed with the Follow-up blood test(ST2) and TTE in OPD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 19 or older
* Patients with acute coronary syndrome who underwent successful percutaneous coronary intervention
* Patients with left ventricular ejection fraction less than 50% on transthoracic echocardiography
* Patients who voluntarily agreed to participate in the study

Exclusion Criteria:

* Failure to obtain TIMI 3 flow after procedure
* If the remaining life span is less than one year
* Women who are breastfeeding or plan to become pregnant or are planning to become pregnant during the study period

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome who underwent successful percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
ST2 and LV end-diastolic volume index | 3 months
  the correlation between changes of ST2 and LV end-diastolic volume index

SECONDARY OUTCOMES:
ST2 and LV ejection fraction | 3 months
  the correlation between changes of ST2 and LV ejection fraction
ST2 and E over e' ratio | 3 months
  the correlation between changes of ST2 and E over e' ratio
ST2 and LV wall motion score | 3 months
  the correlation between changes of ST2 and LV wall motion score

CONTACTS AND LOCATIONS:
Overall Officials: Hyung-Seop Kim, Postdoctoral, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Keimyung University Dongsan Hospital, Daegu, Dalseogu, South Korea